CLINICAL TRIAL: NCT01060878
Title: Phase II, Randomised, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Tolerability of PYM50028 in Subjects With Early-stage Parkinson's Disease Administered Once Daily for 28 Weeks
Brief Title: Investigation of Cogane (PYM50028) in Early-stage Parkinson's Disease (CONFIDENT-PD)
Acronym: CONFIDENT-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phytopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P58/07CL/ST/09/02
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Parkinson's Disease
Keywords: Early-stage
MeSH Terms: conditions — Parkinson Disease | interventions — sarsasapogenin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose I (Experimental)
  Interventions: Drug: PYM50028
- Dose II (Experimental)
  Interventions: Drug: PYM50028
- Dose III (Experimental)
  Interventions: Drug: PYM50028
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PYM50028 — IMP
  Arms: Dose I; Dose II; Dose III
Drug: Placebo — Matching placebo comprising identical vehicle to active doses
  Arms: Placebo

SUMMARY:
A study to test the therapeutic benefit of the compound PYM50028, versus placebo, in treating early-stage Parkinson's disease. Therapeutic benefit will be assessed using the Unified Parkinson's Disease Rating Scale (UPDRS). It is hypothesised that PYM50028 will be safe and well tolerated in this study and demonstrate therapeutic benefit in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of early-stage idiopathic PD within the 2 years prior to screening
* subjects who are not currently receiving any PD treatment

Exclusion Criteria:

* female of child-bearing potential
* history of neurosurgical procedures for PD
* history of severe psychiatric illness

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale parts II & III combined score | 28 Weeks

CONTACTS AND LOCATIONS:
Locations (111):
- United States (41):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Coastal Neurological Medical Group, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Pacific Neuroscience, Oxnard, California
  - Ellison Ambulatory Care Center, Sacramento, California
  - The Parkinson's Institute, Sunnyvale, California
  - Colorado Neurological Institute, Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Hartford Hospital, Manchester, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Neurology Clinical Research Inc, Sunrise, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Elks Rehab - Movement Disorders Center, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center Neuroscience Inst., Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health Center, West Bloomfield, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Atlantic Neuroscience Institute, Morristown, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Weil Medical College of Cornell University, New York, New York
  - Duke Parkinson Center, Durham, North Carolina
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - Neurological Institute, Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Adult Neurology, Charlottesville, Virginia
  - Wisconsin Institute for Neurologic and Sleep Disorders, Milwaukee, Wisconsin
- Canada (8):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - London Health Science Centre, London, Ontario
  - Parkinsons Neurodegenerative Disorder Clinic, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Clinique Sainte-Anne "Memoire et mouvement", Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove Neurologicka klinika, Hradec Králové
  - Fakultni nemocnice Olomouc Neurologicka klinika, Olomouc
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Clintrial s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze Neurologicka klinika, Prague
- France (3):
  - Centre Hospitalier Henri Mondor, Créteil
  - CHRU de Lille, Lille
  - CHU de Toulouse - Hôpital Purpan, Toulouse
- Germany (15):
  - Universitaetsklinikum Wuerzburg Neurologische Klinik und Poliklinik, Bayern
  - Neurologisches Fachkrankenhaus für Bewegungsstörungen / Parkinson, Beelitz-Heilstätten
  - Klinik für Neurologie Charité, Universitaetsmedizin Berlin, Berlin
  - Ruhr-Universität Bochum, Bochum
  - Rheinische Friedrich-Wilhelms-Universität, Bonn
  - Klinikum-Bremerhaven Reinkenheide, Bremerhaven
  - Neurologische Universitätsklinik, Klinikum Carl Gustav Carus, Dresden
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Paracelsus-Elena-Klinik, Kassel
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Gertrudis Klinik Biskirchen, Leun-Biskirchen
  - Neurologische Klinik Lübeck, Lübeck
  - Philipps-Universität Marburg, Marburg
  - Neurologische Klinik und Poliklinik, Klinikum Rechts der Isar TU-Muenchen, Munich
  - Universitätsklinikum Tübingen (UKT), Tübingen
- Hungary (11):
  - Semmelweis Egyetem AOK Neurologiai Klinika, Budapest
  - Fovarosi Onkormanyzat Uzsoki utcai Korhaza Neurologiai Osztaly, Budapest
  - Jahn Ferenc Del-pesti Korhaz Neurologiai Osztaly, Budapest
  - De Oec Áok, Debrecen
  - Kenezy Korhaz Rendelointezet Egeszsegugyi Szolgaltato Nonprofit Korlatolt Felelossegu Tarsasag Neurologiai Osztaly, Debrecen
  - Petz Aladar Megyei Oktato Korhaz Neurologiai Osztaly, Győr
  - Kaposi Mór Oktató Kórház, Kaposvár
  - Bacs-Kiskun Megyei Onkormanyzat Korhaza Neurologiai es Stroke Osztaly, Kecskemét
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Neurologiai Klinika, Szeged
  - Veszprem Megyei Csolnoky Ferenc Korhaz Nonprofit Zrt Ideggyogyaszati es Agyerbetegsegek Osztalya, Veszprém
  - Zala Megyei Korhaz Neurologiai Osztaly, Zalaegerszeg
- Poland (5):
  - NZOZ Medica Pro Familia Sp z o o, Katowice
  - Małopolskie Centrum Medyczne, Krakow
  - Krakowska Akademia Neurologii Sp z o o, Krakow
  - prof nadzw dr hab med Andrzej Bogucki Gabinet Lekarski, Lodz
  - NZOZ Medica Pro Familia Sp z o o, Warsaw
- Romania (5):
  - Cabinet Medical Individual de Neurologie Dr. Falup-Pecurariu G. Cristian-Gavril, Brasov
  - Spitalul Clinic de Recuperare Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Cai Ferate Constanta, Constanța
  - Spitalul Clinic de Urgenta "Prof. Dr. Nicolae Oblu" Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Serbia (4):
  - Klinicko-bolnicki centar "Bezanijska Kosa" Odeljenje za neurologiju i psihijatriju, Belgrade
  - Klinicko-bolnicki centar "Zvezdara" Odeljenje za neurologiju, Belgrade
  - Klinički centar Srbije, Belgrade
  - Kliničko-bolnički centar, Belgrade
- United Kingdom (14):
  - Luton and Dunstable Hospital Foundation Trust, Luton, Bedfordshire
  - Cambridge Centre for Brain Repair, Cambridge, Cambridgeshire
  - The Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - West Suffolk Hospitals NHS Trust, Bury Saint Edmonds, Suffolk
  - Clinical Ageing Research Unit, Newcastle upon Tyne, Tyne and Wear
  - Fairfield General Hospital, Bury
  - Southern General Hospital, Glasgow
  - Walton Centre for Neurology and Neurosurgery, Liverpool
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Charing Cross Hospital, London
  - Salford Royal Foundation Trust, Salford